CLINICAL TRIAL: NCT00511602
Title: Efficacy and Safety of Inhaled Technosphere Insulin Compared to Technosphere Placebo in Patients With Type 2 Diabetes Mellitus Following Diabetes Education
Brief Title: Study of the Efficacy and Safety of Inhaled Technosphere Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDC-INS-0008
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Technosphere Insulin Inhalation Powder (Experimental)
  Interventions: Drug: Technosphere Insulin
- Technosphere Inhalation Powder (Placebo Comparator)
  Interventions: Drug: Technosphere Placebo

INTERVENTIONS:
Drug: Technosphere Insulin — Technosphere Insulin Inhalation Powder
  Arms: Technosphere Insulin Inhalation Powder
Drug: Technosphere Placebo — Technosphere Inhalation Powder
  Arms: Technosphere Inhalation Powder

SUMMARY:
Primary objective to evaluate the effect of a 12-week treatment period with prandial administration of Technosphere Insulin on glucose control in subjects with T2 DM. Secondary objective is to Evaluate the safety and tolerability of a 12-week treatment period of Technosphere Insulin and Technosphere Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2 DM of >2 years and <12 years duration
* Insulin treatment naive treated with diet/exercise or single/combination oral anti-diabetic agents, such as metformin, sulfonylurea, and/or thiazolidinediones
* Stable regimen for >3 months of oral anti-diabetes medication prior to enrollment
* HbA1c >6.6% and <10.5%
* BMI <38 kg/m2
* 18-80 years of age
* Baseline FVC and FEV1 >80% and <120% of predicted normal as measured by spirometry
* Baseline DLCO >80% and <120% of predicted normal

Exclusion Criteria:

* Clinical diagnosis of type 1 diabetes mellitus
* Subjects currently using insulin therapy or at the time of screening
* Known hypersensitivity to the study drug or to drugs of similar chemical structures
* Fasting plasma glucose >270 mg/dL without adequate explanation of a transient causality (screen could be repeated after a 2-week interim period)
* History of severe or multiple allergies
* History of tobacco or nicotine test at screening
* Severe complications of diabetes including history of blindness from or Stage III or IV diabetic retinopathy, history of renal failure requiring dialysis or transplantation, history of amputation of limbs or digits related to diabetic vasculopathy
* Treatment with another investigational drug within 3 months prior to study entry (and for the duration of the study)
* Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids, beta blockers, with the exception of beta blocker ophthalmic solutions for glaucoma or ocular hypertension, or hydrochlorothiazide (HCTZ) at doses >25 mg/day
* Recent loss (within the 2 months prior to screening) of >5% of body weight
* Evidence of moderate or greater ketones in urine or ketoacidosis at screening
* History of chronic obstructive pulmonary disease or history of other known chronic pulmonary disease such as reactive airway disease, chronic bronchitis, emphysema, or asthma
* Diagnosis of AIDS or ARC
* A major psychiatric disorder that would have precluded satisfactory participation in this study
* Subjects who had had a myocardial infarction or stroke within the preceding six months
* Prior diagnosis of systemic autoimmune or collagen vascular disease requiring heart disease graded as Class III or Class IV according to New York Heart Association criteria
* Prior treatment with, or participation in, a clinical study involving an inhaled insulin product
* History of malignancy within 5 years of study entry (other than basal cell carcinoma)
* Significant hepatic disease (as evidenced by ALT or AST >3 times the reference normal range or bilirubin >1.5 times the reference normal range)
* Significant renal disease (as evidenced by creatinine >1.5 mg/dL for males or >1.3 mg/dL for females), proteinuria as evidenced by greater than "small" by dipstick measurement or >2 grams in 24 hours, dialysis, or history of renal transplant
* History of previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2003-12; Primary Completion 2004-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline (week 2) to end of treatment (week 12) | 12 weeks

SECONDARY OUTCOMES:
Area under the plasma glucose concentration versus time (AUCglucose) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after TI administration
Maximum glucose concentration (Cmax) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after TI administration
Time to maximum glucose concentration (tmax) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after TI administration
Area under the plasma glucose concentration versus time (AUCglucose) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after Technosphere Placebo administration
Maximum glucose concentration (Cmax) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after Technosphere Placebo administration
Time to maximum glucose concentration (tmax) | every 4 weeks
  Timepoints: 0, 30, 60, and 120 minutes after Technosphere Placebo administration
Safety variables included adverse events (AEs), clinical laboratory tests, vital signs and physical examinations | every 2 weeks

REFERENCES:
- [Derived] Rosenstock J, Bergenstal R, Defronzo RA, Hirsch IB, Klonoff D, Boss AH, Kramer D, Petrucci R, Yu W, Levy B; 0008 Study Group. Efficacy and safety of Technosphere inhaled insulin compared with Technosphere powder placebo in insulin-naive type 2 diabetes suboptimally controlled with oral agents. Diabetes Care. 2008 Nov;31(11):2177-82. doi: 10.2337/dc08-0315. Epub 2008 Aug 4. PMID 18678610